CLINICAL TRIAL: NCT00354419
Title: A Dose Finding Study of Total Body Irradiation for Conditioning Patients With Severe Aplastic Anemia Transplanted With Umbilical Cord Blood
Brief Title: Cyclophosphamide, Antithymocyte Globulin, and Total-Body Irradiation in Treating Patients With Severe Aplastic Anemia Undergoing Umbilical Cord Blood Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Woolfrey, Ann, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2030.00; NCI-2010-00191
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Whole-Body Irradiation; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Cyclosporine; Cyclosporins; Cord Blood Stem Cell Transplantation; Transplantation; Mycophenolic Acid; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Radiation: total-body irradiation; Drug: cyclophosphamide; Biological: anti-thymocyte globulin; Drug: cyclosporine; Procedure: umbilical cord blood transplantation; Drug: mycophenolate mofetil; Procedure: bone marrow aspiration; Genetic: DNA analysis; Biological: filgrastim

INTERVENTIONS:
Radiation: total-body irradiation — Undergo radiotherapy
  Other Names: TBI
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: cyclosporine — Given IV
  Other Names: 27-400; ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Procedure: umbilical cord blood transplantation — Undergo transplantation
  Other Names: cord blood transplantation; transplantation, umbilical cord blood; UCB transplantation
Drug: mycophenolate mofetil — Given IV or orally
  Other Names: Cellcept; MMF
Procedure: bone marrow aspiration — Correlative study
Genetic: DNA analysis — Correlative study
Biological: filgrastim — Given IV or SC
  Other Names: G-CSF; granulocyte colony-stimulating factor; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor umbilical cord blood stem cell transplant helps stop the growth of abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of total-body irradiation when given together with cyclophosphamide and antithymocyte globulin in treating patients with severe aplastic anemia undergoing umbilical cord blood transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

I. The objective of this study is to determine the lowest dose of total body irradiation combined with cyclophosphamide and antithymocyte globulin that will achieve sustained engraftment in patients with severe aplastic anemia transplanted with unrelated umbilical cord blood.

OUTLINE: This is a dose-escalation study of total-body irradiation (TBI).

MYELOABLATIVE CONDITIONING REGIMEN: Patients receive cyclophosphamide IV on days -7 to -4, -6 to -3, or -5 to -2 and antithymocyte globulin IV on days -6 to -4, -5 to -3, or -4 to -2.

TBI: Patients undergo TBI twice daily on days -3, -2, and/or -1.

UMBILICAL CORD BLOOD TRANSPLANTATION (UCBT): Patients undergo UCBT on day 0. Patients receive filgrastim (G-CSF) IV or subcutaneously beginning on day 1 and continuing until blood counts recover.

GRAFT-VS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive cyclosporine IV or orally (twice daily for patients >= 6 years of age or 3 times daily for patients < 6 years of age) on days -1 to +180 and mycophenolate mofetil IV or orally (twice daily for patients >= 50 kg or 3 times daily for patients < 50 kg) beginning 4 hours after UCBT and continuing until approximately day +0.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Life-threatening marrow failure of nonmalignant etiology meeting two of the three following criteria: granulocytes < 500/mm^3; a corrected reticulocyte count < 1%; platelet count < 20,000/mm^3
* Failure to respond to the best available immunosuppressive treatment protocol by 75 days after initiation of therapy
* Lack of an HLA-identical family member or closely matched (9 or 10 of 10 HLA-locus match) unrelated marrow donor
* DONOR: Unrelated UCB unit matched for at least 4 of 6 loci
* DONOR: Related UCB unit matched for at least 3 of 6 lock
* Selection of the UCB unit(s) will be based upon matching or mismatching at HLA-A, B antigen level and DRB1 allele level typing; while HLA-C antigen/allele and HLA-DQB1 antigen/allele level typing are not considered in the matching criteria, if available each may be used to optimize unit selection
* Multiple UCB units are allowed to provide sufficient cell dose; when multiple units are selected, the following rules apply: a) the UCB unit with the least HLA disparity will be selected first (i.e., selection priority is 6/6 match > 5/6 match > 4/6 match), additional UCB units may be selected to increase cell dose; b) UCB units must be matched to each other for at least 4 of 6 loci; c) each unit must contain at least 1.5 x 10^7 Total Nucleated Cells per kg recipient weight; d) the total cell dose of the combined units must be at least 3.0 x 10^7 Total Nucleated Cells per kg recipient weight

Exclusion Criteria:

* Severe disease other than aplastic anemia that would severely limit the probability of survival during the graft procedure; patients who present with active fungal infections must be treated to resolve this problem before beginning the conditioning regimen
* HIV seropositive patients
* Patients who have developed clonal cytogenetic abnormalities or a myelodysplastic syndrome (these patients will be considered in separate protocols for myelodysplastic syndrome, etc.)
* Patients with paroxysmal nocturnal hemoglobinuria or Fanconi anemia
* Patients > 40 years of age
* Related or unrelated cord blood units with < 1.5 x 10^7 Total Nucleated Cells per kg recipient weight
* Related or unrelated cord blood units without full testing and negative results for hepatitis A, B, C, HIV, HTLV-1, CMV viruses

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Toxicity

SECONDARY OUTCOMES:
Engraftment

CONTACTS AND LOCATIONS:
Overall Officials: Ann Woolfrey, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States